CLINICAL TRIAL: NCT01726907
Title: A Prospective Comparison of Robotic and Endoscopic SMG Resection Via Retroauricular Approach
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Stopped due to failure to recruit appropriate target patients
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2011-0819
Record Dates: First submitted 2012-11-07; First posted 2012-11-15 (Estimated); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: SMG Resection in Comparison to Endoscopic SMG Resection
Keywords: submandibular gland; robotic; endoscopic; face lift; hairline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Robotic SMG resection (Experimental): Robot-assisted SMG resection
  Interventions: Device: Robotic SMG resection
- Endoscopic SMG resection (Active Comparator): Endoscope-assisted SMG resection
  Interventions: Device: Endoscopic SMG resection

INTERVENTIONS:
Device: Robotic SMG resection — The surgical procedure and the considerations for surrounding neurovascular structures were similar to that of the endoscope-assisted SMG resection. The da Vinci surgical system (Intuitive Surgical Inc., Sunnyvale, CA) including a 30° dual channel endoscopic arm and two instrument arms was introduced. The SMG was retracted using the 5-mm Maryland forceps on the left and the dissection was conducted using a 5-mm spatula monopolar cautery or a Harmonic curved shears on the right. A Yankauer suction handled by a bed-side assistant could be used for counter traction of the gland which facilitated the dissection procedure.
  Arms: Robotic SMG resection
Device: Endoscopic SMG resection — An assistant held a 10-mm 30° rigid endoscope allowing the operating surgeon to use both hands. Surgical resection tools such as dissector and Harmonic scalpel (Harmonic Ace 23E®; Johnson & Johnson Medical, Cincinnati, OH, USA) was held in the right hand and a Yankauer suction or a Debakey forcep was held on the left for traction of the SMG. The dissection plane between the capsule of the SMG was conducted under magnified endoscopic view using the the blade of the Harmonic scalpel and the endoscopic dissector. Routine identification of the marginal mandibular branch of the facial nerve was unnecessary in SMG resection, since the dissection plane was always deep to the middle layer of the deep cervical fascia which includes the fascia of the gland. The Wharton's duct, facial artery and vein were ligated using the Harmonic scalpel or vascular clip.
  Arms: Endoscopic SMG resection

SUMMARY:
Traditional transcervical incision of the upper neck is a safe and effective approach for resection of the submandibular gland (SMG). However, external scar at the highly visible area may be a burden for the patients and sometimes may lead to disfiguring hypertrophic scar or keloid. Recently, the investigators reported our surgical technique of 'endoscope-assisted' and 'robot-assisted' SMG resection, which was feasible and showed excellent cosmetic outcomes since the scar was hidden by the auricle and hair. In our previous feasibility study of robot-assisted SMG resection, the investigators proposed that robot-assisted technique may overcome the limitations of endoscopic instruments with rigid and straight nature without articulation and surgical view of two-dimension. In addition, the ergonomically designed operating system was more convenient for the surgeon considering the frequent collision of the endoscopic instruments and reversed hand-eye coordination in endoscope-assisted surgery. However, clinical trial comparing the surgical outcomes of the two techniques has not been reported in the literature.

In this study, the investigators made a prospective comparative study of robot-assisted versus endoscope-assisted SMG resection to determine whether robot-assisted technique has benefits regarding early surgical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as pleomorphic adenoma or chronic sialadenitis from preoperative ultrasound-guided fine needle aspiration biopsy (FNAB)

Exclusion Criteria:

* Past history of neck surgery or radiation
* Possible malignancy expected from FNAB or image study
* Gland with severe adhesion to surrounding tissue on preoperative physical examination

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-02; Primary Completion 2013-02 (Estimated); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
length of incision | expected average opeartion time : 60~90 minutes
  length of incision is measure by a surgical ruler after before skin incision

SECONDARY OUTCOMES:
amount and duration of drainage | on the day of discharge from hospital (expected average period : postoperative 3 days)
  duration of drainage, hospital stay and complications are measured on the day of discharge by the charge doctor
hospital stay | on the day of discharge from hospital (expected average period : postoperative 3 days)
complications | on the day of discharge from hospital (expected average period : postoperative 3 days)

OTHER OUTCOMES:
size of the tumor and SMG | expected average time : 1 week after surgery
  size of the tumor and SMG is measure by the pathologist
cosmetic satisfaction score | 2 months after surgery
  cosmetic satisfaction score is evaluated at the out-patient department during follow up using the questionnaire with scale of 1 (extremely dissatisfied) to 5 (extremely satisfied)

CONTACTS AND LOCATIONS:
Locations (1):
- epartment of Otorhinolaryngology, Yonsei University College of Medicine, Seoul, South Korea